CLINICAL TRIAL: NCT02809560
Title: Detection of Cav1 Calcium Channels in Inflammatory Cells of Asthmatic Children
Acronym: CAVASTHME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11 054 03
Record Dates: First submitted 2016-05-17; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
Keywords: Lymphocytes Th2; Cav1 channels
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthmatic children (Experimental): Induced sputum method using hypertonic serum
  Interventions: Procedure: Induced sputum method using hypertonic serum
- Control children (Sham Comparator): Induced sputum method using hypertonic serum
  Interventions: Procedure: Induced sputum method using hypertonic serum

INTERVENTIONS:
Procedure: Induced sputum method using hypertonic serum — Collection of expectoration in sterile vial, conserved in ice all along the examination

SUMMARY:
Asthma affects about 10% of children and 6% of adults in industrialized countries. Lymphocytes (L) Th2, a T cell population (LT) producing interleukin (IL) -4, 5 and 13 are broadly involved in this pathology in experimental models and in humans. Many studies show that the signaling pathways activated by the commitment of T receiver differ depending LT. The identification of specific signaling pathways links to Th2 offer new therapeutic approaches. Precedent study showed that mouse Th2 selectively expressed related to calcium channels sensitive channels Cav1 voltage, normally found in excitable cells where they are defined as receivers dihydropyridine (DHP).

The goal of the present study is to show the presence of Cav1 channels in inflammatory cells in allergic asthmatics and show overexpression of these channels in the peripheral blood mononuclear cells from asthmatic subjects before and / or after stimulation with the TCR in comparison with controls.

ELIGIBILITY:
Inclusion Criteria:

For Asthmatic children arm :

* Girl not in childbearing potential or taking contraceptive treatment
* Asthma diagnosis in at least 6 months as defined by clinical symptoms (expiratory dyspnea, wheezing, sibilance) and respiratory function (reversibility of VEMS at least 12% after salbutamol administration)
* Allergologic tests positives to airborne allergens : positive prick test and/or specific IgE > 0,35 kU/L for at least one allergen
* Asthma severity between mild to moderate based on Global initiative for asthma classification during more than one month with inhaled corticotherapies +/- long term action beta -mimetic long compounds (salmeterol, formoterol)
* Patient insured with a social security scheme

For control children arm :

* Girl not in childbearing potential or taking contraceptive treatment
* No medical history of asthma
* No medical history of allergy or symptoms of allergy on skin (atopic dermatitis), respiratory tract (rhino-conjunctivitis, asthma) or food allergy

Exclusion Criteria:

For both arms:

* Chronic respiratory pathology : known occlusive or restrictive respiratory syndrome like interstitial lung disease, neuromuscular disease, mucoviscidoses, respiratory tract abnormalities with cough, dyspnea or digital hippocratism.
* History of pulmonary or nose and throat infectious disease during last 4 months
* Parasitic disease non treated during last 3 months
* Dyspnea during the inclusion
* Systemic corticotherapy during the last 3 months before inclusion
* Immunosuppressive therapy during the last 3 months before inclusion
* Diabeta
* Disease causing immune disorder
* Infection during inclusion
* Participation to another study witch implies medical treatment during last 3 months before inclusion

For asthmatic children arm :

* Chronic pulmonary pathology (excluding asthma)
* Asthma exacerbation during inclusion
* VEMS < 70% of normal range or VEMS < 70% of normal range after inhalation of serum (despite salbutamol administration)
* Patient unable to complete pulmonary function testing

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Detection of sequence coding for Cav1 in cells as assessed by reverse transcription polymerase chain reaction | Day 1

SECONDARY OUTCOMES:
Presence of Cav1 channels as assessed by correlation between Cav1 expression and eosinophils in expectoration collection | Day 1
Presence of Cav1 channels as assessed by correlation between Cav1 expression and lymphocytes T in expectoration collection | Day 1
Comparison of CRTH2+ cells in total blood between asthmatic and control group | Day 1
Comparison of Cav1 channels and cytokines Th2 expression between asthmatic and control group before T-Cell receptor stimulation | Day 1
Comparison of Cav1 channels and cytokines Th2 expression between asthmatic and control group after T-Cell receptor stimulation | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: François Brémont, MD, Principal Investigator — Hôpital des Enfants CHU Toulouse

IPD SHARING:
Plan to Share IPD: No